CLINICAL TRIAL: NCT05298644
Title: A Randomized, Double-Blinded, Active Controlled COVID-19 Study to Evaluate The Safety, Tolerability, And Immunogenicity Of Different Doses Of VLA2001 Vaccine, In Children (≥2 To <12 Years)
Brief Title: COVID-19 Paediatric VLA2001-321 Study
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Valneva has contacted regulators to align on potential adjustments to the previously agreed Pediatric Investigational Plan. Valneva has suspended VLA2001 pediatric development, and study VLA2001-321 will not commence.
Sponsor: Valneva Austria GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VLA2001-321
Record Dates: First submitted 2022-03-16; First posted 2022-03-28 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: SARS-CoV-2 Infection
Keywords: VLA2001; SARS-CoV-2 Infection; COVID-19
MeSH Terms: conditions — COVID-19 | interventions — VLA2001 COVID-19 vaccine

STUDY DESIGN:
Intervention Model Description: Sequential Assignment:
  1. st phase: Dose-finding part participants aged ≥5 to <12 years
  2. nd phase: Dose-finding part participants aged ≥2 to <5 years
  3. rd phase: Confirmatory Part participants aged ≥5 to <12 years
  4. th phase: Confirmatory Part participants aged ≥2 to <5 years
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dose finding ≥5 to <12 years (Experimental): on Day 1 and Day 29 either VLA2001 half dose or VLA2001 full dose
  Interventions: Biological: VLA2001
- Dose finding ≥2 to <5 years (Experimental): on Day 1 and Day 29 either VLA2001 half dose or VLA2001 full dose
  Interventions: Biological: VLA2001
- Confirmatory ≥5 to <12 years (Other): Day 1: VLA2001 selected dose (= either VLA2001 half dose or VLA2001 full dose) Day 29: VLA2001 selected dose (= either VLA2001 half dose or VLA2001 full dose) Day 57: Active Comparator
  Interventions: Biological: VLA2001; Drug: Active Comparator
- Confirmatory ≥2 to <5 years (Other): Day 1: Active Comparator Day 29: VLA2001 selected dose (= either VLA2001 half dose or VLA2001 full dose) Day 57: VLA2001 selected dose (= either VLA2001 half dose or VLA2001 full dose)
  Interventions: Biological: VLA2001; Drug: Active Comparator

INTERVENTIONS:
Biological: VLA2001 — whole virus inactivated SARS-CoV-2 vaccine adjuvanted with cytosine phospho-guanine (CpG)1018 in combination with aluminium hydroxide
Drug: Active Comparator — Menactra, Meningococcal (Groups A, C, Y and W-135) Polysaccharide Diphtheria Toxoid Conjugate Vaccine.
  Arms: Confirmatory ≥2 to <5 years; Confirmatory ≥5 to <12 years

SUMMARY:
This is a Randomized, Double-blinded, Active-controlled Study to evaluate the Safety, Tolerability and Immunogenicity of VLA2001 in participants of ≥2 to 12 years.

In total 1720 participants will receive either VLA2001 or active Comparator.

DETAILED DESCRIPTION:
This is a Randomized, Double-blinded, Active-controlled Study to evaluate the Safety, Tolerability and Immunogenicity of VLA2001 in participants of ≥2 to 12 years.

The study will consist of four parts:

* Dose-finding part (participants aged ≥5 to <12 years)
* Dose-finding part (participants aged ≥2 to <5 years)
* Confirmatory part (participants aged ≥5 to <12 years)
* Confirmatory part (participants aged ≥2 to <5 years)

Dose-finding part (participants aged ≥5 to <12 years) Approximately 60 participants will receive 2 intramuscular doses of either half-dose VLA2001 (n=30) or full-dose VLA2001 (n=30) on Days 1 and 29 in a 1:1 ratio.

Dose-finding part (participants aged ≥2 to <5 years) Approximately 60 participants will receive 2 intramuscular doses of either half-dose VLA2001 (n=30) or full-dose VLA2001 (n=30) on Days 1 and 29 in a 1:1 ratio.

Dose-finding part for age group ≥2 to <5 years will be initiated after dose for age group ≥5 to <12 years is confirmed.

Confirmatory Part (participants aged ≥5 to <12 years and ≥2 to <5 years) Overall, approximately 1600 participants aged ≥2 to <12 years will be enrolled. 800 participants aged ≥5 to <12 years and 800 participants aged ≥2 to <5 years will be randomized in 3:1 ratio. In each age group, 600 participants will receive VLA2001, and 200 participants comparator.

Vaccination will start with either 1 intramuscular dose of VLA2001 (selected dose) or comparator vaccine. 28 days later all participants will receive a dose of VLA2001 (selected dose) and 28 days thereafter those who had received the comparator vaccine will receive their second dose with VLA2001 while those who have already received two doses of VLA2001 will receive the comparator vaccine.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent by the participant's legal representative(s), according to local requirements, and written informed assent of the participant, if applicable, prior to any study related procedures.
2. Participants of either gender aged between 2 years and <12 years at screening.
3. Regarding history of Menactra (meningococcal vaccination): only participants <5 years can be included who received no Menactra vaccination. Participants ≥5 years can be included, if at least 4 years have elapsed since the prior dose.
4. Medically stable such that, according to the judgment of the investigator the participant appears likely to be able to remain on study through the end of protocol-specified follow-up.

   • For participants with chronic diseases (such as, asthma, diabetes mellitus, cystic fibrosis, human immunodeficiency virus [HIV] infection), the disease should be stable, defined as not requiring significant change in therapy or hospitalization for worsening disease during the 3 months prior to the expected day of randomization (Visit 1) and as per investigator assessment.
5. Must be able to attend all visits of the study and comply with all study procedures, including daily completion of the e-Diary after each vaccination.
6. Female participants of non-childbearing potential may be enrolled. For this study, non-childbearing potential is defined as pre-menarche.
7. Female participants of childbearing potential (WOCBP) might be enrolled if:

   * have a negative pregnancy test on the day of vaccination,
   * have practiced adequate contraception* or has abstained from all activities that could result in pregnancy for at least 28 days prior to the first injection,
   * have agreed to continue adequate contraception or abstinence through 3 months following the second injection (Phase 2 part) or following the third vaccination (Phase 3 part),
   * are not currently breastfeeding.

Exclusion Criteria:

1. Participant is pregnant or planning to become pregnant within 3 months after study vaccine administration.
2. History of allergy to any component of the vaccine or its excipients.
3. Prior history of allergic or anaphylactic reaction after previous dose of a meningococcal capsular 12 polysaccharide-, diphtheria toxoid- or CRM197-containing vaccine, or to any component of Menactra.
4. Significant infection (e.g., positive SARS-CoV-2 RT-PCR) or other acute illness, including fever >100.4 °F (>38.0 °C) within 2 weeks prior to administration of vaccine.
5. A medical or psychiatric condition that, according to the investigator's judgment, may pose additional risk as a result of participation, interfere with study assessments, interfere with interpretation of results or compromise participant safety.
6. Participants with history of multisystemic-inflammatory syndrome in children (MIS-C).
7. Participated in an interventional clinical study within 28 days prior to Day 1.
8. Received any non-study vaccine within 28 days before or after any dose of vaccine (except for seasonal influenza vaccine, which is permitted within 14 days before or after any dose of vaccine).
9. Thrombocytopenia or any coagulation disorder that would contraindicate intramuscular injection.
10. Severe and uncontrolled ongoing autoimmune or inflammatory disease, history of Guillain-Barre syndrome, or any other demyelinating condition

    Prior/concomitant therapy:
11. Receipt of immunoglobulin or another blood product within the 3 months before expected day of randomization (Visit 1) in this study or those who expect to receive immunoglobulin or another blood product during this study,
12. Immunosuppressive treatment during the course of the study (unless such treatment has to be administered in an emergency situation). Note: Specifically, treatment that can be expected to influence immune response. Such treatment includes, but is not limited to, systemic or high dose inhaled (>800 μg/day of beclomethasone dipropionate or equivalent) corticosteroids, radiation treatment or other immunosuppressive or cytotoxic drugs. Use of inhaled (low dose), intranasal or topical steroids is permitted

    * Glucocorticoids at a dose ≥20 mg/day of prednisone or equivalent given daily or on alternate days for ≥14 consecutive days between randomization and the participant´s schedule
    * Other systemically administered drugs with significant immunosuppressive activity, such as azathioprine, tacrolimus, cyclosporine, methotrexate, or cytotoxic chemotherapy between randomization and the participant´s schedule
13. Prior administration of an investigational or approved CoV vaccine (such as, SARS-CoV-2, SARS CoV, Middle East Respiratory Syndrome CoV) or planned use during the trial.
14. Treatment with investigational or approved agents for prophylaxis against COVID 19 (such as, receipt of SARS-CoV-2 monoclonal antibodies or oral COVID 19 anti-viral agents) within 6 months prior to enrolment.
15. Receipt of any vaccine (licensed or investigational), other than licensed influenza vaccine, within 28 days prior to the expected day of randomization (Visit 1).

    Others:
16. Any member of the study team or sponsor.
17. An immediate family member or household member of the study's personnel.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2023-07-31 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Frequency and severity of solicited local and systemic adverse events (AE) | up to 7 days after each vaccination
Immune response measured after completion of a 2-dose immunization schedule with VLA2001 as determined by the Geometric Mean Titer (GMT) | 2 weeks after completion of a 2-dose immunization schedule
Immune response measured after completion of a 2-dose immunization schedule with VLA2001 as determined by seroconversion rate (SCR) (defined as 4-fold increase from baseline) of SARS-CoV-2-specific neutralising antibodies | 2 weeks after completion of a 2-dose immunization schedule

SECONDARY OUTCOMES:
Frequency, causality and severity of any Adverse Event (AE) | up to Month 12
  Dose Finding Part
Frequency and causality of any serious adverse events (SAEs) | up to Month 12
  Dose Finding Part
Frequency, causality and severity of medically-attended AEs (MAAEs) | up to Month 12
  Dose Finding Part
Frequency, causality and severity of adverse events of special interest (AESIs) | up to Month 12
  Dose Finding Part
Immune response of VLA2001 as determined by the Geometric Mean Titer (GMT) of SARS-CoV-2-specific neutralising antibodies | up to Month 12
  Dose Finding Part
Immune response of VLA2001 as determined by seroconversion rate (SCR) (defined as 4-fold increase from baseline) of SARS-CoV-2-specific neutralising antibodies | up to Month 12
  Dose Finding Part
Immune response of VLA2001 as determined by the Geometric Mean Titer (GMT) of SARS-CoV-2-specific S-protein binding antibodies | up to Month 12
  Dose Finding Part
Immune response of VLA2001 as determined by seroconversion rate (SCR) (defined as 4-fold increase from baseline) of SARS-CoV-2-specific S-protein binding antibodies | up to Month 12
  Dose Finding Part
Frequency and severity of solicited local and systemic adverse events (AEs) | up to 7 days after each vaccination
  Confirmatory Phase
Frequency, causality and severity of any unsolicited adverse event (AE) up to 4 weeks following the immunization with VLA2001 (administered as a first dose) in comparison to the vaccination with the comparator vaccine (administered as a first dose) | up to 4 weeks following immunization
  Confirmatory Phase
Frequency, causality and severity of any adverse event (AE) | up to Month 12
  Confirmatory Phase
Frequency, causality and severity of participants with medically-attended adverse events (MAAEs) | up to Month 12
  Confirmatory Phase
Frequency and causality of any serious adverse events (SAEs) | up to Month 24
  Confirmatory Phase
Frequency, causality and severity of adverse events of special interest (AESIs) including multisystem inflammatory syndrome in children (MISC) | up to Month 24
  Confirmatory Phase
Immune response of VLA2001 as determined by the Geometric Mean Titer (GMT) of SARS-CoV-2-specific neutralising antibodies | up to Month 12
  Confirmatory Phase
Immune response of VLA2001 as determined by seroconversion rate (SCR) (defined as 4-fold increase from baseline) of SARS-CoV-2-specific neutralising antibodies | up to Month 12
  Confirmatory Phase
Immune response of VLA2001 as determined by the Geometric Mean Titer (GMT) of SARS-CoV-2-specific S-protein binding antibodies | up to Month 12
  Confirmatory Phase
Immune response of VLA2001 as determined by seroconversion rate (SCR) (defined as 4-fold increase from baseline) of SARS-CoV-2-specific S-protein binding antibodies | up to Month 12
  Confirmatory Phase
Assessment of T-cell responses from PBMCs in participants after in vitro stimulation with SARS-CoV-2 antigens using e.g. ELISpot or intracellular cytokine staining | up to Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Valneva Clinical Deveopment, Study Chair — Valneva Austria GmbH

IPD SHARING:
Plan to Share IPD: No